CLINICAL TRIAL: NCT03740425
Title: Transfusion Requirements in Transcatheter Aortic Valve Implantation (TRITAVI) Study
Acronym: TRITAVI
Status: Completed | Type: Observational
Sponsor: G. d'Annunzio University (Other)
Collaborators: IRCCS Policlinico S. Donato (Other); University Hospital, Catania (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Hospital Clínico Universitario de Valladolid (Other)
Responsible Party: Principal Investigator, Marco Zimarino, MD, PhD, G. d'Annunzio University
Other Study IDs: TRITAVI18
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Transcatheter Aortic Valve Implantation (TAVI); Blood Transfusion; AKI; Prognosis; Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Blood Transfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Transfusion: Patients requiring blood transfusion after transcatheter aortic valve implantation (TAVI)
  Interventions: Procedure: Blood Transfusion
- No Transfusion: Patients not requiring blood transfusion after transcatheter aortic valve implantation (TAVI)
  Interventions: Procedure: Blood Transfusion

INTERVENTIONS:
Procedure: Blood Transfusion — Blood Transfusion in patients who underwent transcatheter aortic valve implantation (TAVI)

SUMMARY:
Periprocedural bleeding events are frequent during transcatheter aortic valve implantation (TAVI), mainly driven by vascular complications and are associated to a worse prognosis. Therefore, red blood cell (RBC) transfusion is often required, although it is associated with worsened outcomes.

There is no consensus on the optimal transfusion strategy after bleeding. The Transfusion Requirements in Transcatheter Aortic Valve Implantation (TRITAVI) will be a multicenter retrospective registry enrolling consecutive patients who underwent TAVI; the primary aim of the study will be to test whether RBC transfusion is a marker or an independent predictor of adverse events.

DETAILED DESCRIPTION:
Periprocedural bleeding events are frequent during transcatheter aortic valve implantation (TAVI), mainly driven by vascular complications and are associated to a worse prognosis. Therefore, red blood cell (RBC) transfusion is often required, although it is associated with worsened outcomes.

There is no consensus on the optimal transfusion strategy after bleeding: among patients undergoing cardiac surgery, the Transfusion Requirements in Cardiac Surgery (TRICS) III trial documented that a restrictive RBC transfusion strategy (if hemoglobin level was <7.5 g/dl) was noninferior to a liberal approach (if hemoglobin level was <9.5 g/dl) with respect to the composite occurrence of death, myocardial infarction (MI), stroke, or new-onset renal failure with dialysis.

The Transfusion Requirements in Transcatheter Aortic Valve Implantation (TRITAVI) will be a multicenter retrospective registry enrolling consecutive patients who underwent TAVI; the primary aim of the study will be to test whether RBC transfusion is a marker or an independent predictor of adverse events. Patients will be stratified according to their lowest hemoglobin value (>9.5 g/dl, 7.5-9.5 g/dl and <7.5 g/dl) and to whether they received or not periprocedural RBC transfusion.

The primary endpoint will be the 30-day occurrence of major adverse cardiovascular events (MACE), as death, myocardial infarction (MI), stroke, or acute kidney injury (AKI, as absolute increase in serum creatinine ≥0.3 mg/dL [≥26.4 μmol/L] or ≥50% increase ≤72 hours).

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing transcatheter aortic valve implantation (TAVI)

Exclusion Criteria:

* age<18 years

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All-consecutive patients referring at the participants centers undergoing transcatheter aortic valve implantation (TAVI)
Sampling Method: Probability Sample
Enrollment: 3235 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Major adverse cardiovascular events (MACE) | 30 days and end of follow-up (3 years)
  all-cause death, myocardial infarction (MI), stroke, or acute kidney injury (AKI)

SECONDARY OUTCOMES:
Death | 30 days and end of follow-up (3 years)
  all-cause death, cardiovascular death, non cardiovascular death

OTHER OUTCOMES:
Myocardial infarction | 30 days and end of follow-up (3 years)
  Myocardial infarction
acute kidney injury (AKI) | 30 days
  need for dialYsis or increase in serum creatinine ≥0.3 mg/dL [≥26.4 μmol/L] or ≥50% increase ≤72 hours
stroke | 30 days and end of follow-up (3 years)
  stroke or transient ischemic attack (TIA)

CONTACTS AND LOCATIONS:
Overall Officials: Marco Zimarino, MD, PhD, Principal Investigator — G. d'Annunzio University
Locations (1):
- Santissima Annunziata Hospital, Chieti, Italy

IPD SHARING:
Plan to Share IPD: Undecided
Data will be shared only to other Participants Centers

REFERENCES:
- [Result] Mazer CD, Whitlock RP, Fergusson DA, Hall J, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, McGuinness S, Royse A, Carrier FM, Young PJ, Villar JC, Grocott HP, Seeberger MD, Fremes S, Lellouche F, Syed S, Byrne K, Bagshaw SM, Hwang NC, Mehta C, Painter TW, Royse C, Verma S, Hare GMT, Cohen A, Thorpe KE, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Restrictive or Liberal Red-Cell Transfusion for Cardiac Surgery. N Engl J Med. 2017 Nov 30;377(22):2133-2144. doi: 10.1056/NEJMoa1711818. Epub 2017 Nov 12. PMID 29130845
- [Result] Mazer CD, Whitlock RP, Fergusson DA, Belley-Cote E, Connolly K, Khanykin B, Gregory AJ, de Medicis E, Carrier FM, McGuinness S, Young PJ, Byrne K, Villar JC, Royse A, Grocott HP, Seeberger MD, Mehta C, Lellouche F, Hare GMT, Painter TW, Fremes S, Syed S, Bagshaw SM, Hwang NC, Royse C, Hall J, Dai D, Mistry N, Thorpe K, Verma S, Juni P, Shehata N; TRICS Investigators and Perioperative Anesthesia Clinical Trials Group. Six-Month Outcomes after Restrictive or Liberal Transfusion for Cardiac Surgery. N Engl J Med. 2018 Sep 27;379(13):1224-1233. doi: 10.1056/NEJMoa1808561. Epub 2018 Aug 26. PMID 30146969
- [Derived] Radico F, Biancari F, D'Ascenzo F, Saia F, Luzi G, Bedogni F, Amat-Santos IJ, De Marzo V, Dimagli A, Makikallio T, Stabile E, Blasco-Turrion S, Testa L, Barbanti M, Tamburino C, Porto I, Fabiocchi F, Conrotto F, Pelliccia F, Costa G, Stefanini GG, Macchione A, La Torre M, Bendandi F, Juvonen T, Pasceri V, Wanha W, Benedetto U, Miraldi F, Dobrev D, Zimarino M. Red blood cell transfusion and mortality after transcatheter aortic valve implantation via transapical approach: A propensity-matched comparison from the TRITAVI registry. Int J Cardiol Heart Vasc. 2024 Jul 6;53:101460. doi: 10.1016/j.ijcha.2024.101460. eCollection 2024 Aug. PMID 39070183
- [Derived] Zimarino M, Barbanti M, Dangas GD, Testa L, Capodanno D, Stefanini GG, Radico F, Marchioni M, Amat-Santos I, Piva T, Saia F, Reimers B, De Innocentiis C, Picchi A, Toro A, Rodriguez-Gabella T, Nicolini E, Moretti C, Gallina S, Maddestra N, Bedogni F, Tamburino C. Early Adverse Impact of Transfusion After Transcatheter Aortic Valve Replacement: A Propensity-Matched Comparison From the TRITAVI Registry. Circ Cardiovasc Interv. 2020 Dec;13(12):e009026. doi: 10.1161/CIRCINTERVENTIONS.120.009026. Epub 2020 Dec 4. PMID 33272037